CLINICAL TRIAL: NCT06264206
Title: Effect of Immunomodulatory Treatment on IVF Outcomes in Patients With KIRR AA Genotype: a Retrospective Cohort Study With Implications for Personalized Fertility Strategies
Brief Title: Effect of Immunomodulatory Treatment on IVF (in Vitro Fertilization) Outcomes in Patients With KIR AA Genotype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calla IVF Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALLA_IVF_KIR
Record Dates: First submitted 2024-02-12; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Immunomodulatory Drugs; Killer-cell Immunoglobulin-like Receptors (KIRs); KIR Alleles (KIR AA)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KIR AA (Experimental): Patients from arm KIR AA received immunomodulatory treatment, and the pregnancy rate was calculated after this treatment, and compared to the one before the treatment
  Interventions: Diagnostic Test: Killer-cell immunoglobulin-like receptors (KIRs) testing
- KIR BX (No Intervention): Patients from arm KIR BX did not receive immunomodulatory treatment, and the pregnancy rate was calculated and compared with the ones from arm KIRR AA- before and after immunomodulatory treatment

INTERVENTIONS:
Diagnostic Test: Killer-cell immunoglobulin-like receptors (KIRs) testing — patients were tested for KIRs, and based on the divided in the 2 arms. Patient from ARM KIR AA received immunomuodulatorc treatment.
  Other Names: immunomodulatory treatment for KIR AA
  Arms: KIR AA

SUMMARY:
The aim of the study is to investigate the immune cause of recurrent implantation failure (RIF) and the role of immunomodulatory treatment in IVF (in vitro fertilization) patients that have a KIR AA genotype. We compared pregnancy rates in Group KIR AA without immunomodulatory treatment, and pregnancy rates in Group KIR AA with immunomodulatory treatment.

DETAILED DESCRIPTION:
The investigators included patients that underwent an (IVF )in vitro fertilization procedure in CALLA IVF Clinic Oradea - Romania, between 01 January 2022 and 31 December 2023.

Recurrent implantation failure (RIF) impacts 10% of couples undergoing in vitro fertilization (IVF), prompting the exploration of tailored treatments to address underlying causes and enhance implantation rates. Among these causes, maternal immune tolerance toward embryos has garnered significant attention in RIF research, with Killer-cell immunoglobulin-like receptors (KIRs) on natural killer (NK) cells emerging as key players in maternal-fetal immune interactions. The investigation into KIR alleles (KIR AA) in RIF is rooted in the theory that specific KIR-HLA-C combinations may contribute to implantation failures. Recent studies suggest that KIR genotyping could serve as a predictive tool for RIF, potentially enabling personalized approaches in assisted reproductive technology, such as immunomodulatory treatments and tailored embryo transfers.

All couples underwent IVF ovarian stimulation, with various factors documented including age, type of infertility, number of oocytes retrieved, number of embryos produced, pregnancy rate.

A total of 65 patients were enrolled in this study, with 24 patients included in group A, this is the group with KIR AA and 41 patients included in the group B, meaning the group with the KIR Bx Inclusion criteria: patients with an infertility diagnosis having an IVF procedure with at least two top-quality embryo to transfer (according to Gardners criteria), that sign the accord to be enrolled in this study with a negative test for chronic endometritis and normal hysteroscopic findings, also patients that have an history of recurrent pregnancy loss and have an IVF indication will be tested in the first round.

Exclusion criteria: absence of signed consent, refusal of hysteroscopy, uterine abnormalities, thin endometrium, endometrial polyps, pelvic cancer, acute inflammatory disease, Asherman syndrome, chronic endometritis, oocyte or spermatozoa donor.

The KIR AA group experienced improved pregnancy outcomes compared to those in the same cohort who did not undergo prior immunomodulatory treatment

ELIGIBILITY:
Inclusion Criteria:

* patients with an infertility diagnosis having an IVF procedure with at least two top-quality embryo to transfer (according to Gardners criteria)
* patients that sign the accord to be enrolled in this study
* patients with a negative test for chronic endometritis and normal hysteroscopic findings,
* patients that have an history of recurrent pregnancy loss and have an IVF indication will be tested in the first round.

Exclusion Criteria:

* absence of signed consent
* refusal of hysteroscopy
* uterine abnormalities
* thin endometrium
* endometrial polyps
* pelvic cancer
* acute inflammatory disease
* Asherman syndrome
* chronic endometritis

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 65 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
the incidence of immune cause of recurrent implantation failure | 3-6 months
the efficiency of immnomodulatory treatment on pregnancy rate in patients with KIR AA | 3-6 months

SECONDARY OUTCOMES:
comparation between the pregnancy rates in KIR AA group and KIR Bx group | 3-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Calla Ivf Center, Oradea, Bihior, Romania